CLINICAL TRIAL: NCT02076698
Title: Clinical and Medico-economical Assessment of Deep Brain Stimulation of the Anterior Nucleus of the Thalamus for the Treatment of Pharmacoresistant Partial Epilepsy
Brief Title: Deep Brain Stimulation of the Anterior Nucleus of the Thalamus in Epilepsy
Acronym: FRANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1317 FRANCE
Record Dates: First submitted 2014-02-20; First posted 2014-03-03 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Partial Epilepsy; Surgery
Keywords: Deep Brain Stimulation; Anterior Nucleus of thalamus; Treatment refractory; Pharmacoresistant partial epilepsy; vagus nerve stimulation therapy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AN-DBS (Experimental): Deep Brain Stimulation of the Anterior Nucleus of the thalamus
  Interventions: Procedure: AN-DBS
- Usual treatment (Active Comparator): Usual treatment of epilepsy including vagus nerve stimulation (VNS)
  Interventions: Drug: Usual treatment

INTERVENTIONS:
Procedure: AN-DBS — Electrode and one multichannel stimulator surgical time: 4 to 6 hours 3 visits of adjustment
  Other Names: Deep Brain Stimulation
  Arms: AN-DBS
Drug: Usual treatment — usual treatment of epilepsy Vagus nerve stimulation: maintained
  Other Names: Treatment of epilepsy including vagus nerve stimulation
  Arms: Usual treatment

SUMMARY:
The main objective of the study is twofold:

1. Assess the clinical efficacy of DBS on epilepsy according to their number and severity at 1 year follow up.
2. Perform a cost-effectiveness analysis from the perspective of Medicare at 1 and 2 years.

The study hypothesis is that thalamic DBS (neurostimulation of the anterior nucleus of the thalamus) will decrease significantly, the frequency (potentially 50% reduction in severe crises) of the most severe seizures, in at least 50% of patients who have drug-resistant partial epilepsy; and should also improve significantly the quality of life through a gain of independence in activities of daily life, the possible recovery of functional abilities, recovery of social or professional activities.

ELIGIBILITY:
Inclusion Criteria:

* Patient with focal or multifocal epilepsy with or without secondary generalized seizure inoperable at the time of inclusion
* Failure of pharmacological therapies (pharmacoresistant epilepsy) for over 4 years (persistent seizures despite at least two anti-epileptic treatments used at the optimal dose for at least 2 years)
* Failure of vagus nerve stimulation, defined as the persistence of crises considered debilitating after 2 years of VNS's treatment
* VNS failure in a patient treated with VNS, for less than 2 years. with stop early due to the worsening crisis
* Intelligence quotient above 55
* Have the written consent of the legal representative for patients under guardianship and minors
* Affiliation to the french social security system or equivalent
* People who signed the consent form
* Seizure frequency at least 4 crisis / month on average for at least 3 months, about 12 crisis in 3 months objectified by the neurologist during visit pre-inclusion, and confirmed by the neurologist after 3 months of Baseline during the inclusion visit

Exclusion Criteria:

* Patient with a generalized epilepsy Immediately
* Patient with a simple partial seizures (subjective manifestations only)
* Patient with a cons-indication for MRI, a serious intercurrent disease, a progressive brain tumor
* Patient with a suicide risk of in the six months preceding the inclusion visit (score ≥ 2 on item 10 of the Montgomery-Asberg Depression Rating Scale)
* Patient a surgical or anesthetic cons-indication
* Patient with anticoagulant or antiplatelet treatment in the long term
* Woman of childbearing potential without effective contraception, or pregnant or lactating
* People hospitalized without consent
* People deprived of freedom
* Patient currently participating in another clinical research, or who participated in a clinical study in the month preceding the pre-inclusion visit (except for any non-interventional research)

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Assessment of effectiveness of thalamic DBS on seizures severity | 2 years
  The main objective of the study is twofold : to assess the effectiveness of DBS on seizures according to their severity at 1 year follow up and to perform a cost-effectiveness analysis from the perspective of Medicare at 1 and 2 years.

SECONDARY OUTCOMES:
Cost-utility analysis from the perspective of Medicare | 2 years
  Perform a cost-utility analysis from the perspective of Medicare at 1 and 2 years.
Comparison of the improvement of quality of life and overall neuropsychological impact | 2 years
  Compare the improvement of quality of life and overall neuropsychological impact at 1 and 2 years.
Comparison the adverse effects (including depression) | 2 years
  Compare the adverse events (special focus on depression) at 1 and 2 years.
Impact of th new therapeutic strategy on the hospital budget | 2 years
  Determine the impact on the hospital budget for the introduction of this therapeutic strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan CHABARDES, MDPHD, Principal Investigator — University Hospital, Grenoble
Locations (12):
- France (12):
  - University Hospital of Pellegrin, Bordeaux
  - University Hospital of Grenoble Michallon, Grenoble
  - University Hospital, Lille
  - University Hospital of Pierre Wertheimer, Lyon
  - University Hospital of la Timone, Marseille
  - University Hospital of Gui de Chauliac, Montpellier
  - University Hospital, Nancy
  - University Hospital Pasteur, Nice
  - Sainte Anne Hospital, Paris
  - University Hospital of La Pitié-Salpétrière, Paris
  - University Hospital of Pontchaillou, Rennes
  - University Hospital of Rangueil, Toulouse

REFERENCES:
- [Background] Chabardes S, Kahane P, Minotti L, Koudsie A, Hirsch E, Benabid AL. Deep brain stimulation in epilepsy with particular reference to the subthalamic nucleus. Epileptic Disord. 2002 Dec;4 Suppl 3:S83-93. PMID 12495878
- [Background] Chabardes S, Minotti L, Chassagnon S, Piallat B, Torres N, Seigneuret E, Vercueil L, Carron R, Hirsch E, Kahane P, Benabid AL. [Basal ganglia deep-brain stimulation for treatment of drug-resistant epilepsy: review and current data]. Neurochirurgie. 2008 May;54(3):436-40. doi: 10.1016/j.neuchi.2008.02.039. Epub 2008 May 2. French. PMID 18452956
- [Background] Fisher R, Salanova V, Witt T, Worth R, Henry T, Gross R, Oommen K, Osorio I, Nazzaro J, Labar D, Kaplitt M, Sperling M, Sandok E, Neal J, Handforth A, Stern J, DeSalles A, Chung S, Shetter A, Bergen D, Bakay R, Henderson J, French J, Baltuch G, Rosenfeld W, Youkilis A, Marks W, Garcia P, Barbaro N, Fountain N, Bazil C, Goodman R, McKhann G, Babu Krishnamurthy K, Papavassiliou S, Epstein C, Pollard J, Tonder L, Grebin J, Coffey R, Graves N; SANTE Study Group. Electrical stimulation of the anterior nucleus of thalamus for treatment of refractory epilepsy. Epilepsia. 2010 May;51(5):899-908. doi: 10.1111/j.1528-1167.2010.02536.x. Epub 2010 Mar 17. PMID 20331461
- [Background] Lim SN, Lee ST, Tsai YT, Chen IA, Tu PH, Chen JL, Chang HW, Su YC, Wu T. Electrical stimulation of the anterior nucleus of the thalamus for intractable epilepsy: a long-term follow-up study. Epilepsia. 2007 Feb;48(2):342-7. doi: 10.1111/j.1528-1167.2006.00898.x. PMID 17295629